CLINICAL TRIAL: NCT01764945
Title: Relative Bioavailability of BI 201335 (Capsule) Compared to Three Different Oral Solutions of BI 201335 Following Oral Administration in Healthy Male and Female Volunteers (an Open-label, Randomised, Single-dose, Four-way Crossover Study)
Brief Title: Relative Bioavailability of BI 201335 Capsule Versus Three Different Oral Solutions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1220.46; 2012-000687-22 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
MeSH Terms: interventions — faldaprevir

ARMS (2):
- 1 BI 201335 (Experimental): low dose
  Interventions: Drug: BI 201335 (Reference); Drug: BI 201335 (Test)
- 2 BI 201335 (Experimental): high dose
  Interventions: Drug: BI 201335 (Test); Drug: BI 201335 (Reference)

INTERVENTIONS:
Drug: BI 201335 (Reference) — soft gelatine capsule, oral administration
  Arms: 1 BI 201335
Drug: BI 201335 (Test) — oral solution 3
  Arms: 1 BI 201335
Drug: BI 201335 (Test) — oral solution 3
  Arms: 2 BI 201335
Drug: BI 201335 (Test) — oral solution 2
  Arms: 1 BI 201335
Drug: BI 201335 (Reference) — soft gelatine capsule, oral administration
  Arms: 2 BI 201335
Drug: BI 201335 (Test) — oral solution 1
  Arms: 2 BI 201335
Drug: BI 201335 (Test) — oral solution 1
  Arms: 1 BI 201335
Drug: BI 201335 (Test) — oral solution 2
  Arms: 2 BI 201335

SUMMARY:
The objective of the current study is to investigate the relative bioavailability of two different doses of BI 201335, administered as soft gelatine capsule in comparison to the equivalent doses of three different oral solution per dose of BI 201335.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects

Exclusion criteria:

Any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1220.46.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- 40mg Faldaprevir: Sequence Group ADBC: 40 mg group: The reference treatment was a single 40 mg dose of faldaprevir soft gelatine capsule (treatment A) and the test treatments were single 40 mg doses of 3 different faldaprevir oral solutions (treatments B, C, and D).
  The order of treatment administration in this sequence group is ADBC with washout phases of at least 14 days between drug administrations.
  Oral administration (under fed conditions, i.e. following a high-fat breakfast).
- 40mg Faldaprevir: Sequence Group BACD: 40 mg group: The reference treatment was a single 40 mg dose of faldaprevir soft gelatine capsule (treatment A) and the test treatments were single 40 mg doses of 3 different faldaprevir oral solutions (treatments B, C, and D).
  The order of treatment administration in this sequence group is BACD with washout phases of at least 14 days between drug administrations.
  Oral administration (under fed conditions, i.e. following a high-fat breakfast).
- 40mg Faldaprevir: Sequence Group CBDA: 40 mg group: The reference treatment was a single 40 mg dose of faldaprevir soft gelatine capsule (treatment A) and the test treatments were single 40 mg doses of 3 different faldaprevir oral solutions (treatments B, C, and D).
  The order of treatment administration in this sequence group is CBDA with washout phases of at least 14 days between drug administrations.
  Oral administration (under fed conditions, i.e. following a high-fat breakfast).
- 40mg Faldaprevir: Sequence Group DCAB: 40 mg group: The reference treatment was a single 40 mg dose of faldaprevir soft gelatine capsule (treatment A) and the test treatments were single 40 mg doses of 3 different faldaprevir oral solutions (treatments B, C, and D).
  The order of treatment administration in this sequence group is DCAB with washout phases of at least 14 days between drug administrations.
  Oral administration (under fed conditions, i.e. following a high-fat breakfast).
- 120mg Faldaprevir: Sequence Group EHFG: 120 mg group: The reference treatment was a single 120 mg dose (consisting of three 40 mg faldaprevir soft gelatine capsules, treatment E) and the test treatments were single 120 mg doses of 3 different faldaprevir oral solutions (treatments F, G, and H).
  The order of treatment administration in this sequence group is EHFG with washout phases of at least 14 days between drug administrations.
  Oral administration (under fed conditions, i.e. following a high-fat breakfast).
- 120mg Faldaprevir: Sequence Group FEGH: 120 mg group: The reference treatment was a single 120 mg dose (consisting of three 40 mg faldaprevir soft gelatine capsules, treatment E) and the test treatments were single 120 mg doses of 3 different faldaprevir oral solutions (treatments F, G, and H).
  The order of treatment administration in this sequence group is FEGH with washout phases of at least 14 days between drug administrations.
  Oral administration (under fed conditions, i.e. following a high-fat breakfast).
- 120mg Faldaprevir: Sequence Group GFHE: 120 mg group: The reference treatment was a single 120 mg dose (consisting of three 40 mg faldaprevir soft gelatine capsules, treatment E) and the test treatments were single 120 mg doses of 3 different faldaprevir oral solutions (treatments F, G, and H).
  The order of treatment administration in this sequence group is GFHE with washout phases of at least 14 days between drug administrations.
  Oral administration (under fed conditions, i.e. following a high-fat breakfast).
- 120mg Faldaprevir: Sequence Group HGEF: 120 mg group: The reference treatment was a single 120 mg dose (consisting of three 40 mg faldaprevir soft gelatine capsules, treatment E) and the test treatments were single 120 mg doses of 3 different faldaprevir oral solutions (treatments F, G, and H).
  The order of treatment administration in this sequence group is HGEF with washout phases of at least 14 days between drug administrations.
  Oral administration (under fed conditions, i.e. following a high-fat breakfast).
Period: Overall Study
Arm/Group | 40mg Faldaprevir: Sequence Group ADBC | 40mg Faldaprevir: Sequence Group BACD | 40mg Faldaprevir: Sequence Group CBDA | 40mg Faldaprevir: Sequence Group DCAB | 120mg Faldaprevir: Sequence Group EHFG | 120mg Faldaprevir: Sequence Group FEGH | 120mg Faldaprevir: Sequence Group GFHE | 120mg Faldaprevir: Sequence Group HGEF
Started | 5 | 5 | 5 | 5 | 10 | 8 | 9 | 9
Completed | 5 | 4 | 5 | 5 | 10 | 8 | 8 | 9
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: This trial was an open-label study consisting of two (40mg and 120mg Faldaprevir) 4-way crossover groups. All subjects were to receive 4 treatments: either treatments A, B, C, and D (20 subjects) or treatments E, F, G, and H (36 subjects). Subjects were randomised to 1 of the 4 treatment sequences for each dose group to be tested in a 1:1:1:1 ratio
Groups:
- Total: Total of all reporting groups
Arm/Group | 40mg Faldaprevir: Sequence Group ADBC | 40mg Faldaprevir: Sequence Group BACD | 40mg Faldaprevir: Sequence Group CBDA | 40mg Faldaprevir: Sequence Group DCAB | 120mg Faldaprevir: Sequence Group EHFG | 120mg Faldaprevir: Sequence Group FEGH | 120mg Faldaprevir: Sequence Group GFHE | 120mg Faldaprevir: Sequence Group HGEF | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 10 | 8 | 9 | 9 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (5.3) | 39.8 (5.1) | 38.0 (10.2) | 44.4 (4.2) | 33.9 (9.7) | 38.6 (9.6) | 39.4 (8.1) | 34.9 (9.5) | 38.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 2 | 5 | 4 | 7 | 3 | 28
  Male | 3 | 2 | 3 | 3 | 5 | 4 | 2 | 6 | 28

OUTCOME MEASURES:

1. Primary Outcome: AUC0-∞
Description: Area under the concentration-time curve of the analyte (faldaprevir) in plasma over the time interval from 0 extrapolated to infinity.
  The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: -1:00, 1:00, 2:00, 3:00, 4:00, 5:00, 6:00, 7:00, 8:00, 9:00, 10:00, 12:00, 24:00, 48:00, 72:00, 96:00, 120:00 h (hours) after administration of faldaprevir on Day 1.
Population: Pharmacokinetic analysis set (PK set) includes all subjects who provided evaluable data for at least 1 evaluable observation for a PK endpoint in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- 40mg Faldaprevir: Treatment A: 40 mg faldaprevir soft gelatine capsule (reference).
- 40mg Faldaprevir: Treatment B: 40 mg faldaprevir oral solution 1
- 40mg Faldaprevir: Treatment C: 40 mg faldaprevir oral solution 2
- 40mg Faldaprevir: Treatment D: 40 mg faldaprevir oral solution 3
- 120mg Faldaprevir: Treatment E: 120 mg faldaprevir soft gelatine capsule (reference).
- 120mg Faldaprevir: Treatment F: 120 mg faldaprevir oral solution 1
- 120mg Faldaprevir: Treatment G: 120 mg faldaprevir oral solution 2
- 120mg Faldaprevir: Treatment H: 120 mg faldaprevir oral solution 3
Arm/Group | 40mg Faldaprevir: Treatment A | 40mg Faldaprevir: Treatment B | 40mg Faldaprevir: Treatment C | 40mg Faldaprevir: Treatment D | 120mg Faldaprevir: Treatment E | 120mg Faldaprevir: Treatment F | 120mg Faldaprevir: Treatment G | 120mg Faldaprevir: Treatment H
Number analyzed (Participants) | 19 | 19 | 20 | 18 | 35 | 35 | 36 | 35
ng*h/mL | 3960 (32.3) | 3400 (28.5) | 3350 (28.4) | 3420 (30.4) | 15000 (34.5) | 13900 (38.8) | 14500 (38.3) | 14100 (36.0)
Statistical Analysis 1: Comparison: 40mg Faldaprevir: Treatment A vs 40mg Faldaprevir: Treatment B; relative bioavailability comparison of 40 mg faldaprevir soft gelatine capsules compared with the equivalent dose of an oral solution. (treatment B : treatment A); Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 82.58, 90% CI 2-sided [73.69 to 92.54], Standard Deviation 19.7 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: 40mg Faldaprevir: Treatment A vs 40mg Faldaprevir: Treatment C; relative bioavailability comparison of 40 mg faldaprevir soft gelatine capsules compared with the equivalent dose of an oral solution. (treatment C : treatment A); Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 83.34, 90% CI 2-sided [73.65 to 94.30], Standard Deviation 22.2 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 3: Comparison: 40mg Faldaprevir: Treatment A vs 40mg Faldaprevir: Treatment D; relative bioavailability comparison of 40 mg faldaprevir soft gelatine capsules compared with the equivalent dose of an oral solution. (treatment D : treatment A); Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 83.92, 90% CI 2-sided [74.69 to 94.28], Standard Deviation 19.6 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 4: Comparison: 120mg Faldaprevir: Treatment E vs 120mg Faldaprevir: Treatment F; relative bioavailability comparison of 120 mg faldaprevir soft gelatine capsules compared with the equivalent dose of an oral solution. (treatment F : treatment E); Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 92.90, 90% CI 2-sided [88.94 to 97.04], Standard Deviation 10.5 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 5: Comparison: 120mg Faldaprevir: Treatment E vs 120mg Faldaprevir: Treatment G; relative bioavailability comparison of 120 mg faldaprevir soft gelatine capsules compared with the equivalent dose of an oral solution. (treatment G : treatment E); Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 96.37, 90% CI 2-sided [91.55 to 101.43], Standard Deviation 12.7 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 6: Comparison: 120mg Faldaprevir: Treatment E vs 120mg Faldaprevir: Treatment H; relative bioavailability comparison of 120 mg faldaprevir soft gelatine capsules compared with the equivalent dose of an oral solution. (treatment H : treatment E); Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 94.44, 90% CI 2-sided [89.88 to 99.24], Standard Deviation 12.0 — the standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Cmax
Description: Maximum measured concentration of the analyte (faldaprevir) in plasma. The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: -1:00, 1:00, 2:00, 3:00, 4:00, 5:00, 6:00, 7:00, 8:00, 9:00, 10:00, 12:00, 24:00, 48:00, 72:00, 96:00, 120:00 h after administration of faldaprevir on Day 1.
Population: PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 40mg Faldaprevir: Treatment A | 40mg Faldaprevir: Treatment B | 40mg Faldaprevir: Treatment C | 40mg Faldaprevir: Treatment D | 120mg Faldaprevir: Treatment E | 120mg Faldaprevir: Treatment F | 120mg Faldaprevir: Treatment G | 120mg Faldaprevir: Treatment H
Number analyzed (Participants) | 19 | 19 | 20 | 18 | 35 | 35 | 36 | 35
ng/mL | 86.4 (36.0) | 65.4 (39.0) | 64.0 (40.4) | 69.7 (28.1) | 625.0 (47.3) | 481.0 (47.1) | 488.0 (52.1) | 485.0 (48.4)
Statistical Analysis 1: Comparison: 40mg Faldaprevir: Treatment A vs 40mg Faldaprevir: Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 74.07, 90% CI 2-sided [65.44 to 83.83], Standard Deviation 21.5 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: 40mg Faldaprevir: Treatment A vs 40mg Faldaprevir: Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 73.23, 90% CI 2-sided [63.33 to 84.68], Standard Deviation 26.2 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 3: Comparison: 40mg Faldaprevir: Treatment A vs 40mg Faldaprevir: Treatment D; [analysis description as in outcome 1, analysis 3]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 78.76, 90% CI 2-sided [68.94 to 89.99], Standard Deviation 22.7 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 4: Comparison: 120mg Faldaprevir: Treatment E vs 120mg Faldaprevir: Treatment F; [analysis description as in outcome 1, analysis 4]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 78.30, 90% CI 2-sided [71.42 to 85.84], Standard Deviation 22.5 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 5: Comparison: 120mg Faldaprevir: Treatment E vs 120mg Faldaprevir: Treatment G; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 78.43, 90% CI 2-sided [69.54 to 88.46], Standard Deviation 30.4 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 6: Comparison: 120mg Faldaprevir: Treatment E vs 120mg Faldaprevir: Treatment H; [analysis description as in outcome 1, analysis 6]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 78.09, 90% CI 2-sided [69.35 to 87.94], Standard Deviation 29.4 — the standard deviation is actually the geometric coefficient of variation

3. Primary Outcome: AUC0-tz
Description: Area under the concentration-time curve of the analyte (faldaprevir) in plasma over the time interval from 0 to the time of the last quantifiable data point.
  The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 2
Population: PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 40mg Faldaprevir: Treatment A | 40mg Faldaprevir: Treatment B | 40mg Faldaprevir: Treatment C | 40mg Faldaprevir: Treatment D | 120mg Faldaprevir: Treatment E | 120mg Faldaprevir: Treatment F | 120mg Faldaprevir: Treatment G | 120mg Faldaprevir: Treatment H
Number analyzed (Participants) | 19 | 19 | 20 | 18 | 35 | 35 | 36 | 35
ng*h/mL | 3020 (29.4) | 2600 (32.9) | 2520 (38.3) | 2550 (34.3) | 14200 (35.2) | 12900 (39.4) | 13400 (38.0) | 13100 (37.0)
Statistical Analysis 1: Comparison: 40mg Faldaprevir: Treatment A vs 40mg Faldaprevir: Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 82.02, 90% CI 2-sided [75.98 to 88.55], Standard Deviation 13.1 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: 40mg Faldaprevir: Treatment A vs 40mg Faldaprevir: Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 80.93, 90% CI 2-sided [74.58 to 87.83], Standard Deviation 14.5 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 3: Comparison: 40mg Faldaprevir: Treatment A vs 40mg Faldaprevir: Treatment D; [analysis description as in outcome 1, analysis 3]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 79.60, 90% CI 2-sided [74.84 to 84.67], Standard Deviation 10.2 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 4: Comparison: 120mg Faldaprevir: Treatment E vs 120mg Faldaprevir: Treatment F; [analysis description as in outcome 1, analysis 4]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 91.59, 90% CI 2-sided [87.53 to 95.84], Standard Deviation 11.0 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 5: Comparison: 120mg Faldaprevir: Treatment E vs 120mg Faldaprevir: Treatment G; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 94.38, 90% CI 2-sided [89.76 to 99.24], Standard Deviation 12.4 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 6: Comparison: 120mg Faldaprevir: Treatment E vs 120mg Faldaprevir: Treatment H; [analysis description as in outcome 1, analysis 6]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 92.91, 90% CI 2-sided [88.42 to 97.63], Standard Deviation 12.0 — the standard deviation is actually the geometric coefficient of variation

ADVERSE EVENTS:
Time Frame: AEs and concomitant medication will be evaluated continuously from first drug administration until the end-of-study examination (up to 5 weeks). AEs persisting after trial completion must be followed up, until they have normalised.
Description: Subjects were required to report spontaneously any AEs throughout the clinical trial. In addition, each volunteer was assessed regularly by the medical staff throughout the clinical trial as well as at the end of observation and whenever necessary as deemed by the investigator.
Arm/Group | 40mg Faldaprevir: Treatment A | 40mg Faldaprevir: Treatment B | 40mg Faldaprevir: Treatment C | 40mg Faldaprevir: Treatment D | 120mg Faldaprevir: Treatment E | 120mg Faldaprevir: Treatment F | 120mg Faldaprevir: Treatment G | 120mg Faldaprevir: Treatment H
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/20 | 0/19 | 0/35 | 0/36 | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 3/19 | 2/20 | 8/20 | 6/19 | 6/35 | 5/36 | 7/36 | 8/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 40mg Faldaprevir: Treatment A (N=19) | 40mg Faldaprevir: Treatment B (N=20) | 40mg Faldaprevir: Treatment C (N=20) | 40mg Faldaprevir: Treatment D (N=19) | 120mg Faldaprevir: Treatment E (N=35) | 120mg Faldaprevir: Treatment F (N=36) | 120mg Faldaprevir: Treatment G (N=36) | 120mg Faldaprevir: Treatment H (N=35)
Oral herpes (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 4 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 4 | 1 | 1 | 3 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.